CLINICAL TRIAL: NCT01370070
Title: Multicenter Phase II Study of MK-2206 in Previously Treated Patients With Recurrent and Metastatic Nasopharyngeal Carcinoma
Brief Title: MK-2206 in Recurrent Nasopharyngeal Carcinoma
Acronym: MC1079
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Cancer Trial Units, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC024
Record Dates: First submitted 2011-05-12; First posted 2011-06-09 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — MK 2206

ARMS (1):
- MK-2206 (Experimental)
  Interventions: Drug: MK-2206

INTERVENTIONS:
Drug: MK-2206 — 200mg weekly repeated q 28 days

SUMMARY:
To evaluate the activity and safety of MK-2206 in patients with recurrent or metastatic nasopharyngeal carcinoma (NPC)

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 year, able to give written informed consent.
* History of histologically or cytologically confirmed non-keratinizing NPC that has recurred at locoregional and/or distant sites, and is not amenable to potentially curative radiotherapy or surgery.
* Patients must have progressed within 24 months of receiving one or two prior line of chemotherapy for recurrent disease, of which at least one line must contain platinum drugs such as Cisplatin, Carboplatin or oxaliplatin.
* Adequate organ reserve: neutrophils >1.5x109/L, platelets ≥100 x109/L, hemoglobin ≥9 g/dL, serum alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) or ALT< 5 x ULN in the presence of liver metastases, serum bilirubin < 2.5 x ULN, serum creatinine < 1.5 x ULN.
* Presence of measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST ver 1.1).

Exclusion Criteria:

* Chemotherapy, radiotherapy (except to bone metastases) or investigational treatment within 4 weeks of enrollment.
* Patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled before the patient enters the trial.
* Cardiovascular: baseline QTcF > 450 msec (male) or QTcF >470 msec (female) Left bundle branch block, 2nd or 3rd degree AV block, bifascicular block, sick sinus syndrome, Wolff-Parkinson-white syndrome, significant sinus bradycardia (< 50bpm) . However, patients with asymptomatic right bundle branch block or 1st degree AV block, in the absence of known cardiac disease (e.g. coronary, valvular) are NOT excluded..
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients alive and progression-free at 6 months along with the confirmed response rate as a dual primary endpoint | 3 years

SECONDARY OUTCOMES:
Adverse events | 2 Years
Overall survival | 3 years
Progression-free survival | 3 Years
RECIST-based subjective response | 3 Years
Laboratory correlates: pharmacokinetics, plasma EBV DNA half-life | 3 years
treatment tolerability | 2 years
duration of response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Ma, MD, FRACP, Principal Investigator — Department of Clinical Oncology, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ma BB, Goh BC, Lim WT, Hui EP, Tan EH, Lopes Gde L, Lo KW, Li L, Loong H, Foster NR, Erlichman C, King AD, Kam MK, Leung SF, Chan KC, Chan AT. Multicenter phase II study of the AKT inhibitor MK-2206 in recurrent or metastatic nasopharyngeal carcinoma from patients in the mayo phase II consortium and the cancer therapeutics research group (MC1079). Invest New Drugs. 2015 Aug;33(4):985-91. doi: 10.1007/s10637-015-0264-0. Epub 2015 Jun 19. PMID 26084990